CLINICAL TRIAL: NCT01243034
Title: Variability of Waist Circumference Measurements at 3 Sites and Its Relationship With Cardiovascular Risk Factors in Patients With Schizophrenia
Brief Title: Waist Circumference Measurements in Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Chen Chang, attending psychiatrist, Changhua Christian Hospital
Other Study IDs: 100717
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Waist Circumference Measurements; Schizophrenia; Cardiovascular Risk Factor
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of metabolic syndrome(MS) among pt's with schizophrenia has been reported to be high, ranging from 24 to 43% in males and 27 to 52% in females. Schizophrenic patients with MS have an increased incidence of DM, coronary heart disease and increased mortality from cardiovascular diseases. Central adiposity is highly correlated with the presence of hypertension, coronary heart disease, type 2 diabetes, and increased mortality risk. Waist circumference(WC) is a better indicator of abdominal obesity and a better predictor of CVD than either BMI or waist-to-hip ratio. However, currently there is no standard location for the measurement of WC.

Objectives: 1. To compare the magnitude of WC measured at 3 sites ( immediately above the iliac crest, midpoint between the lowest rib and the iliac crest , umbilical level) in males and females.

2. To examine the correlation of WC with Triglyceride, cholesterol, HDL, LDL and glucose.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with schizophrenia or schizoaffective disorder (DSM-IV 295) age 18 till 65 years old.

  * Body weight change less than 1 kg in previous one month before index date.

Exclusion Criteria:

* • Patients with a previous hyperlipidemia diagnosis or antilipemic prescription during the preceding 30 days.

  * Patients received any anti-hypertensives or oral hypoglycemic agents.
  * Pregnant or breast-feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: schizophrenia outpatients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2011-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan